CLINICAL TRIAL: NCT03628287
Title: Program Refinements to Optimize Model Impact and Scalability Based on Evidence
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Denis Nash, Professor, City University of New York, School of Public Health
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH117793 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hiv
Keywords: viral load suppression; medical case management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design: To compare effects of the original and revised CCP contemporaneously for timely viral suppression, we will randomize (within matched pairs and one trio) 17 veteran CCP-implementing agencies to immediate or delayed implementation of the revised model, with delayed implementers providing services under the original model until their assigned start date 9 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Original Care Coordination Program (Active Comparator): Specific intervention components include: 1) outreach for initial case finding and after any missed appointment; 2) case management, including social services and benefits assessments; 3) multidisciplinary care team communication and decision-making via case conferences; 4) patient navigation, including appointment reminders, assistance with scheduling appointments, transportation resources, and accompaniment to primary care visits; 5) antiretroviral treatment adherence support, including directly observed therapy for individuals with greatest need; and 6) structured health promotion, for which clients are assigned to program tracks (determining their frequency of health promotion visits: weekly, monthly or quarterly), depending on their level of assessed need.
  Interventions: Other: Original Care Coordination Program
- Revised Care Coordination Program (Experimental): The revised model includes the original intervention components without program track assignments or the three-month induction period of weekly visits. Program additions include a set of tools for assessment and counseling around client HIV self-management capacity; allowance of video chat for delivery of some services; and optional "immediate" antiretroviral therapy (iART: ensuring the client has a filled prescription within 4 days of enrollment or diagnosis). Other changes include greater guidance on recruiting individuals with unsuppressed VL and a switch from per-member-per-day reimbursement to fee-for-service reimbursement that accounts for resource demands, such as staff travel to clients' homes, and offers higher rates for meeting performance standards.
  Interventions: Other: Revised Care Coordination Program

INTERVENTIONS:
Other: Revised Care Coordination Program — Greater focusing, tailoring and cues for delivery of key components of Care Coordination
  Arms: Revised Care Coordination Program
Other: Original Care Coordination Program — Original Care Coordination
  Arms: Original Care Coordination Program

SUMMARY:
In New York, the achievement of 90-90-90 goals is jeopardized not by limited access to affordable care and treatment, but by persistent disparities in HIV viral suppression (VS). Complex behavioral and structural barriers to achieving and maintaining VS require coordinated, combination approaches to meet medical and social service needs. In 2009, at 28 Ryan White Part A (RWPA)-funded agencies, the New York City (NYC) Department of Health and Mental Hygiene (DOHMH) launched a multi-component HIV Care Coordination Program (CCP) directed toward the most vulnerable persons living with HIV (PLWH) in NYC. A systematic CCP effectiveness study began in 2013 (R01 MH101028; PIs: Irvine, Nash). Findings to date suggest that the CCP is superior to usual care for vulnerable subgroups of PLWH, but there remains substantial room for improvement in short- and long-term VS. In an immediate evidence-to-practice feedback loop, the DOHMH is implementing a refined CCP model in 2018. Greater focusing, tailoring and cues for delivery of key components are expected to increase CCP engagement, reach, fidelity, scalability, effectiveness and impact. The aim of the proposed study is to estimate the effect of the revised (vs. original) CCP on timely VS (within 4 months of enrollment), using experimental methods.

DETAILED DESCRIPTION:
Stepped-wedge design. The 17 veteran CCP implementers re-awarded to provide RWPA Care Coordination services in 2018 will be randomized to immediate or delayed implementation of the revised CCP model, with delayed implementers continuing to provide services under the original model until their assigned start date 9 months later, so that we can rigorously and contemporaneously compare effects of the original and revised CCP for the outcome of timely VS. The outcome measure will be derived from the New York City HIV surveillance registry, a population-based data source of longitudinal laboratory (VL, CD4) testing records on all diagnosed NYC PLWH, regardless of medical provider within NYC, and for periods extending before and after program enrollment or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* The original CCP permits enrollment of HIV-infected adults or emancipated minors who are eligible for local Ryan White Part A services (based on residence in the NYC grant area and a household income <435% of federal poverty level) and are 1) newly HIV-diagnosed; 2) out of care >9 months or never in care; 3) missing visits or irregularly in care; 4) exhibiting high VL, VL rebound, or antiretroviral therapy (ART) resistance; 5) new to ART; 6) incompletely adherent to ART; or 7) facing a potential barrier to adherence
* The revised CCP permits enrollment of HIV-infected adults or emancipated minors who are eligible for local Ryan White Part A services (based on residence in the NYC grant area and a household income <435% of federal poverty level) and are 1) newly HIV-diagnosed; 2) out of care >9 months or never in care; 3) virally unsuppressed at the most recent known viral load test in the past 12 months; 4) living with untreated hepatitis C; 5) pregnant; 6)undergoing a change in ART regimen or 7)experiencing other high risk for falling out of medical care or becoming unsuppressed. For criteria (6) and (7), eligibility is conditional upon Self-management Assessment results, unless additional criteria are met.

Exclusion Criteria:

* The stepped-wedge experiment is limited to HIV patients who are virally unsuppressed at the time of program enrollment. Individuals with VL <200 copies/mL at last test before or on the day of program enrollment will be excluded from the comparison of model effects on timely viral suppression (TVS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nash, PhD, Principal Investigator — CUNY School of Public Health and Health Policy; Mary Irvine, DrPH, Principal Investigator — New York City Department of Health and Mental Hygiene
Locations (17):
- United States (17):
  - HHC Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center - STAR Health Center, Brooklyn, New York
  - Sunset Park Health Council, Inc., Brooklyn, New York
  - Wyckoff Heights Medical Center, Brooklyn, New York
  - HHC Elmhurst Hospital Center, Elmhurst, New York
  - Mount Sinai- Beth Israel Medical Center, New York, New York
  - Housing Works Inc, New York, New York
  - Callen Lorde Community Health Center, New York, New York
  - APICHA Community Health Center, New York, New York
  - Mount Sinai-St. Luke's - Roosevelt Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - The Institute for Family Health, New York, New York
  - Services for the Underserved, Inc., New York, New York
  - Community Health Action Of Staten Island, Staten Island, New York
  - Bronx Lebanon Hospital Center, The Bronx, New York
  - Argus Community Inc, The Bronx, New York
  - HHC Jacobi Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
Due to the legal restrictions (New York Public Health Law Article 21, Title III) and the confidential nature of HIV surveillance data in New York, public health authorities in New York City cannot release individual-level data on reported HIV cases for purposes other than ensuring appropriate HIV care. The NYC DOHMH staff are available to assist external researchers who may have further specific data questions or uses. Please send an email to hivreport@health.nyc.gov with questions or requests for additional information.

REFERENCES:
- [Background] Robertson MM, Waldron L, Robbins RS, Chamberlin S, Penrose K, Levin B, Kulkarni S, Braunstein SL, Irvine MK, Nash D. Using Registry Data to Construct a Comparison Group for Programmatic Effectiveness Evaluation: The New York City HIV Care Coordination Program. Am J Epidemiol. 2018 Sep 1;187(9):1980-1989. doi: 10.1093/aje/kwy103. PMID 29788080
- [Background] Irvine MK, Chamberlin SA, Robbins RS, Kulkarni SG, Robertson MM, Nash D. Come as You Are: Improving Care Engagement and Viral Load Suppression Among HIV Care Coordination Clients with Lower Mental Health Functioning, Unstable Housing, and Hard Drug Use. AIDS Behav. 2017 Jun;21(6):1572-1579. doi: 10.1007/s10461-016-1460-4. PMID 27342990
- [Background] Irvine MK, Chamberlin SA, Robbins RS, Myers JE, Braunstein SL, Mitts BJ, Harriman GA, Laraque F, Nash D. Improvements in HIV care engagement and viral load suppression following enrollment in a comprehensive HIV care coordination program. Clin Infect Dis. 2015 Jan 15;60(2):298-310. doi: 10.1093/cid/ciu783. Epub 2014 Oct 9. PMID 25301208
- [Background] Robertson MM, Penrose K, Irvine MK, Robbins RS, Kulkarni S, Braunstein SL, Waldron L, Harriman G, Nash D. Impact of an HIV Care Coordination Program on Durable Viral Suppression. J Acquir Immune Defic Syndr. 2019 Jan 1;80(1):46-55. doi: 10.1097/QAI.0000000000001877. PMID 30299346
- [Background] Nash D, Robertson MM, Penrose K, Chamberlin S, Robbins RS, Braunstein SL, Myers JE, Abraham B, Kulkarni S, Waldron L, Levin B, Irvine MK. Short-term effectiveness of HIV care coordination among persons with recent HIV diagnosis or history of poor HIV outcomes. PLoS One. 2018 Sep 24;13(9):e0204017. doi: 10.1371/journal.pone.0204017. eCollection 2018. PMID 30248136
- [Background] Penrose K, Robertson M, Nash D, Harriman G, Irvine M. Social Vulnerabilities and Reported Discrimination in Health Care Among HIV-Positive Medical Case Management Clients in New York City. Stigma Health. 2020 May;5(2):179-187. doi: 10.1037/sah0000187. Epub 2019 Aug 12. PMID 32432165
- [Background] Stevens ER, Nucifora KA, Irvine MK, Penrose K, Robertson M, Kulkarni S, Robbins R, Abraham B, Nash D, Braithwaite RS. Cost-effectiveness of HIV care coordination scale-up among persons at high risk for sub-optimal HIV care outcomes. PLoS One. 2019 Apr 25;14(4):e0215965. doi: 10.1371/journal.pone.0215965. eCollection 2019. PMID 31022280
- [Derived] Hernandez M, Guarino H, Kozlowski S, Srivastava A, Schenkel R, Tapia T, Seabrook TB, Nash D, Irvine MK. Addressing Mental Health Barriers in HIV Care Coordination Is Crucial to Providing Optimal HIV/AIDS Care. AIDS Patient Care STDS. 2024 Mar;38(3):107-114. doi: 10.1089/apc.2023.0240. PMID 38471091
- [Derived] Irvine MK, Levin B, Abdelqader F, Carmona J, Avoundjian T, Thomas J, Braunstein SL, Robertson M, Nash D. Evaluation of the Revised Versus Original Ryan White Part A HIV Care Coordination Program in a Cluster-Randomized, Stepped-Wedge Trial. J Acquir Immune Defic Syndr. 2023 Apr 1;92(4):325-333. doi: 10.1097/QAI.0000000000003139. Epub 2022 Dec 22. PMID 36729538
- [Derived] Irvine MK, Levin B, Robertson MM, Penrose K, Carmona J, Harriman G, Braunstein SL, Nash D. PROMISE (Program Refinements to Optimize Model Impact and Scalability based on Evidence): a cluster-randomised, stepped-wedge trial assessing effectiveness of the revised versus original Ryan White Part A HIV Care Coordination Programme for patients with barriers to treatment in the USA. BMJ Open. 2020 Jul 27;10(7):e034624. doi: 10.1136/bmjopen-2019-034624. PMID 32718922

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Older New York City HIV surveillance registry datasets were used to determine trial eligibility for the original protocol, excluding clients who died during follow-up. 16 clients who died within 4 months of Care Coordination Program (CCP) or revised-CCP enrollment were added as eligible for trial outcome analyses. Updated surveillance and match datasets identified additional eligible individuals based on latest reported viral load at time of CCP or revised-CCP enrollment, who were also included.
Groups:
- Early-implementation: Early-implementing sites received the revised intervention starting in August 2018 (start of Period 1), with follow-up through January 2020 (end of Period 2).
- Later-implementation: Later-implementing sites received the revised intervention starting in May 2019 (start of Period 2), with follow-up through January 2020 (end of Period 2).
Period: Overall Study
Arm/Group | Early-implementation | Later-implementation
Started | 531 | 429
Period 0: No Revised Program Delivery ((November 2017-March 2018, follow-up through July 2018)) | 83 | 93
Period 1: Revised Program Delivery Only at Sites Assigned to Early Implementation ((August-December 2018, follow-up through April 2019)) | 286 | 104
Period 2: Revised Program Delivery at All Sites ((May-September 2019, follow-up through January 2020)) | 162 | 232
Completed | 531 | 429
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-implementation | Later-implementation | Total
Number analyzed (Participants) | 531 | 429 | 960
Age, Customized [Count of Participants; unit: Participants]
  <25 years | 24 | 32 | 56
  Between 25 and 44 years | 194 | 205 | 399
  Between 45 and 54 years | 148 | 90 | 238
  >=55 years | 165 | 102 | 267
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender man or boy | 331 | 295 | 626
  Cisgender woman or girl | 185 | 112 | 297
  Identified as transgender, gender nonconforming, non-binary, or not sure/questioning (TGNCNB) | 15 | 22 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 183 | 146 | 329
  Not Hispanic or Latino | 347 | 283 | 630
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian/Pacific Islander | 0 | 15 | 15
  Black or African American | 318 | 230 | 548
  White | 24 | 25 | 49
  More than one race/Other | 5 | 13 | 18
  Unknown or Not Reported | 1 | 0 | 1
  Hispanic or Latino | 183 | 146 | 329
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Bronx | 244 | 97 | 341
  United States: Brooklyn | 147 | 173 | 320
  United States: Manhattan | 82 | 72 | 154
  United States: Queens | 24 | 71 | 95
  United States: Staten Island | 22 | 7 | 29
  United States: Outside NYC but within NY EMA | 2 | 5 | 7
  United States: Unknown | 10 | 4 | 14
Primary Language [Count of Participants; unit: Participants]
  English | 437 | 304 | 741
  Other | 94 | 124 | 218
  Unknown | 0 | 1 | 1
Country of Birth [Count of Participants; unit: Participants]
  US/US territory | 433 | 237 | 670
  Other country | 98 | 192 | 290
Transmission Risk [Count of Participants; unit: Participants]
  Men who have sex with men (MSM) | 149 | 172 | 321
  Injection drug users (IDU) | 32 | 18 | 50
  MSM/IDU | 3 | 5 | 8
  Heterosexual | 298 | 207 | 505
  Perinatal | 32 | 20 | 52
  Other/Unknown | 17 | 7 | 24
Housing Status [Count of Participants; unit: Participants]
  Stably housed | 378 | 351 | 729
  Unstably housed or unhoused | 153 | 78 | 231
Incarceration History [Count of Participants; unit: Participants]
  Never | 352 | 355 | 707
  Last 12 months | 25 | 10 | 35
  >12 months ago | 147 | 61 | 208
  Unknown | 7 | 3 | 10
Sexual Orientation [Count of Participants; unit: Participants] — Self-reported; 'other' includes clients who identified their sexual orientation as queer, pansexual, not sure/questioning, or other.
  Participants
    Gay or Lesbian | 125 | 141 | 266
    Straight or Heterosexual | 339 | 240 | 579
    Bisexual | 33 | 31 | 64
    Other/Unknown | 34 | 17 | 51
Mental Health Diagnosis/Condition [Count of Participants; unit: Participants]
  Yes | 286 | 147 | 433
  No | 222 | 259 | 481
  Unknown | 23 | 23 | 46
Recent Hard Drug Use [Count of Participants; unit: Participants] — Hard drug use refers to the use of cocaine/crack, heroin, crystal meth, or prescription drugs to get high.
  Participants
    Yes | 113 | 70 | 183
    No | 407 | 354 | 761
    Unknown | 11 | 5 | 16
Lifetime Hard Drug Use [Count of Participants; unit: Participants] — Hard drug use refers to the use of cocaine/crack, heroin, crystal meth, or prescription drugs to get high.
  Participants
    Yes | 178 | 116 | 294
    No | 343 | 309 | 652
    Unknown | 10 | 4 | 14
Insurance Status [Count of Participants; unit: Participants]
  Insured | 476 | 299 | 775
  Uninsured | 55 | 130 | 185
Employment Status [Count of Participants; unit: Participants]
  Any paid employment | 76 | 134 | 210
  No paid employment | 451 | 283 | 734
  Unknown | 4 | 12 | 16
Federal Poverty Level (FPL) [Count of Participants; unit: Participants]
  <100% of FPL | 456 | 324 | 780
  100%-200% of FPL | 54 | 78 | 132
  >200% of FPL | 21 | 27 | 48
Educational Level [Count of Participants; unit: Participants]
  ≤High school/GED or equivalent | 398 | 302 | 700
  >High school/GED | 130 | 124 | 254
  Unknown | 3 | 3 | 6
Time Since Diagnosis [Count of Participants; unit: Participants]
  ≤1 year pre-enrollment | 51 | 103 | 154
  >1 to 10 years pre-enrollment | 111 | 110 | 221
  >10 to 20 years pre-enrollment | 199 | 114 | 313
  >20 years pre-enrollment | 170 | 102 | 272
Antiretroviral Therapy (ART) Status [Count of Participants; unit: Participants]
  On ART | 479 | 381 | 860
  Not on ART | 52 | 48 | 100
Viral Load [Count of Participants; unit: Participants] — Copies/mL; Eligible participants with no viral load test result at the time of their enrollment were classified as unsuppressed.
  Participants
    200-1,499 | 101 | 80 | 181
    1,500-9,999 | 85 | 74 | 159
    10,000+ | 339 | 264 | 603
    No viral load at enrollment | 6 | 11 | 17
Cluster of differentiation 4 (CD4) Count [Count of Participants; unit: Participants]
  <200 | 234 | 188 | 422
  200-499 | 196 | 156 | 352
  500+ | 94 | 76 | 170
  No CD4 at enrollment | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Timely Viral Suppression (TVS)
Description: TVS defined as achieving viral suppression (VL <200 copies/mL) on the last VL test in the four months following CCP enrollment.
Time Frame: Four months after CCP enrollment
Population: The final analysis used an intention-to-treat design and included all 960 participants recruited at baseline. No participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Early-implementation | Later-implementation
Number analyzed (Participants) | 531 | 429
Participants
  Achieved TVS (suppressed within four months) | 254 | 261
  Did not achieve TVS (unsuppressed) | 277 | 168

ADVERSE EVENTS:
Time Frame: The five-month enrollment periods were: November 2017 through March 2018 (Period 0, with TVS follow-up through July 2018), August through December 2018 (Period 1, with follow-up through April 2019), and May through September 2019 (Period 2, with follow-up through January 2020). For TVS outcome follow-up, each client was followed for 4 months from their specific CCP or revised-CCP enrollment date. Clients were not followed for adverse outcomes beyond a client's specific 4-month follow-up period.
Description: Adverse event definitions did not differ from clinicaltrials.gov definitions.
Arm/Group | Early-implementation | Later-implementation
All-Cause Mortality (participants affected / at risk) | 9/531 | 7/429
Serious Adverse Events (participants affected / at risk) | 0/531 | 0/429
Other Adverse Events (participants affected / at risk) | 0/531 | 0/429

LIMITATIONS AND CAVEATS:
This was an observational trial. The only change made for the purpose of this trial was randomization (within matched pairs) of sites to early or delayed implementation of program revisions. No test, data collection, or treatment was administered specifically for this trial. All persons observed were enrolling for HIV Care Coordination regardless of the trial, and all received the original or revised model of Care Coordination, based on the site and period in which they joined the program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03628287/Prot_SAP_000.pdf